CLINICAL TRIAL: NCT03987802
Title: An Indian Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Post Marketing Surveillance Study of Fiasp® to Evaluate Safety and Effectiveness in Patients With Diabetes Mellitus in Routine Clinical Practice
Brief Title: An Indian Post Marketing Study of Mealtime Insulin, Fiasp®, to Evaluate Its Safety and Effectiveness in Patients With Diabetes Mellitus in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1218-4489; U1111-1222-9492 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fiasp®: Adult patients with diabetes mellitus (type 1 and type 2) under routine clinical practice in India.
  Interventions: Drug: Faster-acting insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Faster-acting insulin aspart given as subcutaneous (s.c., under the skin) injections according to routine clinical practice. The decision to initiate treatment with commercially available Fiasp® must be made by the patient and the treating physician before and independently from the decision to include the patient in this study.

SUMMARY:
This study is to investigate the effects of Fiasp®, a mealtime insulin, in patients with diabetes mellitus. The purpose of this study is to collect information about Fiasp®, which is prescribed to the participants by their doctors. Participants will administer Fiasp® as prescribed by their doctors. The study will last for about 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, age equal to or above 18 years at the time of signing the informed consent.
* Patients diagnosed with diabetes mellitus.
* Patients scheduled to start treatment with Fiasp® based on the clinical judgement of their treating physician.

Exclusion Criteria:

* Known or suspected hypersensitivity to study product(s) or related products.
* Patients on or likely to use insulin pump therapy during the study period
* Previous participation in this study. Participation is defined as having given signed informed consent.
* Mental incapacity, unwillingness or language barriers hindering adequate understanding or cooperation.
* Participation in any clinical study of an approved or non-approved investigational medicinal product within 1 month before treatment start.
* Any disorder which in the opinion of the treating physician may jeopardise the patient's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diabetes mellitus (type 1 and type 2) under routine clinical practice in India.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Number of events

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs) | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Number of events
Adverse Drug Reactions (ADRs) | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Number of events
Serious Adverse Drug Reactions (SADRs) | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Number of events
Patient reported severe hypoglycaemia | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Episodes/person-year
Patient reported Blood Glucose (BG) confirmed (below 56 mg/dl) hypoglycaemia | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Episodes/person-year
Patient reported Severe or BG confirmed (below 56 mg/dl) hypoglycaemia | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Episodes/person-year
Change in HbA1c | From start of treatment (Week 0) to End of Study Visit (Week 26)
  Percent point (%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (26):
- India (26):
  - Vijayratna Diagnostic & Scientific Obesity Clinic, Ahmedabad, Gujarat
  - Life Care Clinic & Research Centre, Bangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - Aster Medcity, Kochi, Kerala
  - Kerala Institute of Medical Sciences, Trivandrum, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - Zandra Healthcare Pvt Ltd, Mumbai, Maharashtra
  - Apollo Hospital, Navi Mumbai, Mumbai, Maharashtra
  - chelleram Diabetes Institute, Pune, Maharashtra
  - Siddhi Hospital And Laparoscopy Center Pvt Ltd, Pune, Maharashtra
  - Max Super Speciality Hospital, Saket, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Khurda, Odisha
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Max Super Speciality Hospital, Mohali, Mohali, Punjab
  - Santokba Durlabhji Memorial Hospital, Jaipur, Rajasthan
  - Kg Hospital and Post Graduate Medical Institute, Coimbatore, Tamil Nadu
  - Arthur Asirvatham hospital,, Madurai, Tamil Nadu
  - Max Super Speciality Hospital, Ghaziabad, Ghaziabad, Uttar Pradesh
  - Regency Hospital, Kanpur, Uttar Pradesh
  - Medanta Lucknow Hospital, Lucknow, Uttar Pradesh
  - AMRI Hospitals, Dhakuria, Kolkata, West Bengal
  - Apollo Multispeciality Hospital, Kolkata, Kolkata, West Bengal
  - Dr B L Kapur Memorial Hospital, New Delhi
  - Sir Ganga Ram Hospital-Cardiology, New Delhi
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com